CLINICAL TRIAL: NCT04124120
Title: Randomized Comparison of the Outcomes of Single vs Multiple Arterial Grafts in Women (ROMA:Women) Trial
Brief Title: Comparison of the Outcomes of Single vs Multiple Arterial Grafts in Women
Acronym: ROMA:Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York Presbyterian Hospital (Other); Sunnybrook Health Sciences Centre (Other); Cedars-Sinai Medical Center (Other); Columbia University (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1703018094-ROMA-Women
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Heart Diseases; Coronary Artery Disease; Coronary Artery Bypass Grafting
MeSH Terms: conditions — Heart Diseases; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients undergoing coronary artery bypass surgery will be in one of two groups. One group will receive a single arterial graft and the second group will receive two or more arterial grafts.
Who Masked: Outcomes Assessor
Masking Description: The endpoint assessors will be blinded to treatment allocation (PROBE).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Arterial Graft (SAG) group (Experimental): Patients in this group will receive a single arterial graft which will be the left internal thoracic artery. Additional grafts used in this group will all be venous grafts.
  Interventions: Procedure: Single arterial graft
- Multiple Arterial Graft (MAG) group (Experimental): Patients in the group will receive multiple arterial grafts. All patients will receive at least two arterial grafts, the left internal thoracic artery with the addition of either the right internal thoracic artery or the radial artery as the second conduit. Some patients may receive additional arterial grafts consisting of the radial artery, the right internal thoracic artery, or the right gastroepiploic artery.
  Interventions: Procedure: Multiple arterial grafting

INTERVENTIONS:
Procedure: Single arterial graft — This interventions consists of patients receiving the left internal thoracic artery to the left anterior descending coronary artery of the heart. In addition to the left internal thoracic artery patients will receive venous grafts for all additional grafting.
  Arms: Single Arterial Graft (SAG) group
Procedure: Multiple arterial grafting — This intervention consists of the patient receiving the left internal thoracic artery to the left anterior descending coronary artery of the heart. The second arterial graft (right internal thoracic artery or radial artery) will be directed to the major branch of the circumflex. Additional grafts will include saphenous veins or arterial conduits.
  Arms: Multiple Arterial Graft (MAG) group

SUMMARY:
The central hypothesis of ROMA:Women is that the use of multiple arterial grafting (MAG) will improve clinical outcomes and quality of life (QOL) compared to single arterial grafting (SAG).

The specific aims of ROMA:Women are:

Aim 1: Determine the impact of MAG vs SAG on major adverse cardiac and cerebrovascular events in women undergoing coronary artery bypass grafting (CABG). The investigators will compare major adverse cardiac and cerebrovascular events (death, stroke, non-procedural myocardial infarction, repeat revascularization, and hospital readmission for acute coronary syndrome or heart failure) in a cohort of 2,300 women randomized 1:1 to MAG or SAG. Differences by important clinical and surgical subgroups (patients younger or older than 70 years, diabetics, racial and ethnic minorities, on vs off pump CABG, type of arterial grafts used) will also be evaluated. The women enrolled in the ongoing ROMA trial (anticipated to be approximately 690) will be included in ROMA:Women, increasing efficiency and reducing enrollment time.

Hypothesis 1.0. MAG will reduce the incidence of major adverse cardiac and cerebrovascular events.

Hypothesis 1.1. The improvement with MAG will be consistent across key subgroups.

Aim 2: Determine the impact of MAG vs SAG on generic and disease-specific QOL, physical and mental health symptoms in women undergoing CABG. The investigators will compare generic (SF-12, EQ-5D) and disease-specific (Seattle Angina Questionnaire) QOL and physical and mental health symptoms (PROMIS-29) in a sub-cohort of 500 women randomized 1:1 to MAG or SAG (including those enrolled in ROMA:QOL). Differences by important subgroups (as defined above) will also be evaluated.

Hypothesis 2.0. MAG will improve generic and disease-specific QOL compared to SAG.

Hypothesis 2.1. MAG will improve physical and mental health symptoms compared to SAG.

Hypothesis 2.2. The improvement with MAG will be consistent across key subgroups.

DETAILED DESCRIPTION:
ROMA:Women will leverage the infrastructure and the existing women population of the ROMA trial. ROMA:Women has two key Aims. In Aim 1, the investigators will compare major adverse cardiac and cerebrovascular events (death, stroke, non-procedural myocardial infarction, repeat revascularization and hospital readmission for acute coronary syndrome or heart failure) in a cohort of 2,300 women randomized 1:1 to MAG or SAG. In Aim 2, the investigators will compare generic (SF-12, EQ-5D) and disease-specific (Seattle Angina Questionnaire) QOL and physical and mental health symptoms (PROMIS-29) in a sub-cohort of 500 women randomized 1:1 to MAG or SAG. Differences by important subgroups (patients younger or older than 70 years, diabetics, racial and ethnic minorities, on vs off pump CABG, type of arterial grafts used) will also be evaluated.

ROMA:Women is a two-arm, international, multi-center, randomized clinical trial nested in the ROMA trial. ROMA:Women will include all the women enrolled in the parent ROMA trial and will leverage the existing ROMA infrastructure including clinical trial unit, database, case report forms (CRF), randomization system, site training resources, informed consent forms (ICF), regulatory approvals, Central Events Review Committee (CEC) processes/personnel, network of participating sites, site PIs, and study coordinators. The planned randomization procedure, interventions and treatment arms, outcome assessments and follow-up protocol of ROMA:Women are identical to those of the currently ongoing parent ROMA trial. The sites participating in ROMA will continue enrollment of women after the completion of the ROMA trial and additional sites will also be opened to reach the target sample size of ROMA:Women.

ELIGIBILITY:
Inclusion Criteria:

1. Women patients ≥18 years old.
2. Isolated coronary artery bypass grafting.
3. Primary (first time) cardiac surgery procedure.
4. Significant disease of the left main coronary artery or of the left anterior descending and the circumflex coronary system with or without disease of the right coronary artery.

Exclusion Criteria:

* Male gender
* Single graft
* Emergency operation
* Myocardial infarction within 72 hours of surgery
* Left ventricular ejection fraction < 35%
* Any concomitant cardiac or non-cardiac procedure
* Previous cardiac surgery
* Preoperative severe end-organ dysfunction (dialysis, liver failure, respiratory failure), cancer or any co-morbidity that reduces life expectancy to less than 5 years.
* Inability to use the saphenous vein or to use both radial and right internal thoracic arteries
* Anticipated need for coronary thrombo-endarterectomy
* Planned hybrid revascularization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 2300 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Primary outcome for aim 1: Death from any cause, any stroke, non-procedural myocardial infarction, repeat revascularization and hospital readmission for acute coronary syndrome or heart failure. | Postoperatively, minimum 2.5 year follow-up
  The primary outcome for aim 1 will be a composite of the first occurrence of death from any cause, any stroke, non-procedural myocardial infarction (>48 hours after surgery), repeat revascularization and hospital readmission for acute coronary syndrome or heart failure.
Primary outcome for aim 2: Disease-specific quality of life | Postoperatively, minimum 2.5 year follow-up
  Assessed using the Seattle Angina Questionnaire (SAQ), a validated 19-item questionnaire that measures five domains related to coronary disease: angina frequency, physical limitations, quality of life, angina stability, and treatment satisfaction. Scores range from 0 to 100 with higher scores indicating fewer symptoms and better health status. The minimum clinically important difference on the SAQ is 5 points.
  The primary endpoint for aim 2 is the absolute change in the Seattle Angina Questionnaire (SAQ) at 12 months compared to baseline.

SECONDARY OUTCOMES:
Death from any cause, any stroke, non-procedural myocardial infarction, and repeat revascularization. | Postoperatively, minimum 2.5 year follow-up
  One of the secondary outcomes for aim 1: It will be a composite of the first occurrence of death from any cause, any stroke, non-procedural myocardial infarction (>48 hours after surgery), and repeat revascularization.
  This is the primary outcome of the parent ROMA trial.
Death from cardiac cause, any stroke, non-procedural myocardial infarction, repeat revascularization and hospital readmission for acute coronary syndrome or heart failure. | Postoperatively, minimum 2.5 year follow-up
  Another secondary outcome for aim 1: It will be a composite of the first occurrence of death from cardiac cause, any stroke, non-procedural myocardial infarction (>48 hours after surgery), repeat revascularization, and hospital readmission for acute coronary syndrome or heart failure.
Death from any cause | Postoperatively, minimum 2.5 year follow-up
  Another secondary outcome for aim 1: Death will be considered to be cardiac unless a definite non-cardiac cause is identified.
Stroke | Postoperatively, minimum 2.5 year follow-up
  Another secondary outcome for aim 1: Based on the American Heart Association/American Stroke Association Expert Consensus stroke definition, stroke will be identified in case of:
  1. pathological, imaging, or other objective evidence of cerebral ischemic injury in a defined vascular distribution; OR
  2. clinical evidence of cerebral ischemic injury based on symptoms persisting ≥24 hours or until death, and other etiologies excluded.
Non-procedural myocardial infarction | > 48 hours postoperatively, minimum 2.5 year follow-up
  Another secondary outcome for aim 1: Based on the 4th Universal Definition, non-periprocedural myocardial infarction will be identified in case of detection of rise and/or fall of cardiac biomarkers with at least one value above the 99th percentile of the upper reference limit together with evidence of myocardial ischemia with at least one of the following:
  1. symptoms of ischemia
  2. electrocardiogram changes indicative of new ischemia (new ST-T changes or new left bundle branch block)
  3. development of pathological Q waves in the electrocardiogram
  4. imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.
Repeat revascularization | Postoperatively, minimum 2.5 year follow-up
  Another secondary outcome for aim 1: Repeat revascularization will include any percutaneous or surgical revascularization on a grafted coronary artery after the initial operation.
Readmission for acute coronary syndrome | Postoperatively, minimum 2.5 year follow-up
  Another secondary outcome for aim 1: Prolonged ischemic symptoms at rest (usually ≥10 minutes in duration), or accelerating pattern of chest pain that occurs with a lower activity threshold (CCS class III or IV) considered to be myocardial ischemia upon final diagnosis resulting in an unscheduled visit to a healthcare facility resulting in an overnight stay generally within 24 hours of the most recent symptoms, cardiac biomarkers not meeting MI criteria, and ECG or angiographic evidence of ischemia.
Readmission for heart failure | Postoperatively, minimum 2.5 year follow-up
  Another secondary outcome for aim 1: While patients may have multiple simultaneous disease processes, for the outcome event of heart failure requiring hospitalization, the diagnosis of congestive heart failure would need to be the primary process. Heart failure (HF) requiring hospitalization is defined as an event that meets the following criteria:
  i. Requires hospitalization AND ii. Clinical symptoms of heart failure AND iii. Physical signs of heart failure AND iv. Need for additional/increased therapy AND v. No other non-cardiac etiology (such as chronic obstructive pulmonary disease, hepatic cirrhosis, acute renal failure, or venous insufficiency) and no other cardiac etiology (such as pulmonary embolus, cor pulmonale, primary pulmonary hypertension, or congenital heart disease) for signs or symptoms are identified.
Generic quality of life according to the Short Form Health Survey (SF-12v2) | Postoperatively, minimum 2.5 year follow-up
  Secondary outcomes for aim 2: The SF-12v12 measures eight dimensions of health: physical functioning, role limitations due to physical problems, bodily pain, vitality, general health perception, social function, role limitations due to emotional problems, and mental health. Scores for each domain range from 0 to 100 with higher scores indicating better health status.
  The SF-12v2 has two summary measures: physical and mental self-perceived health with norm-based methods that standardize the score to a mean of 50 and standard deviation of 10.
Generic quality of life according to EuroQuol-5D (EQ-5D) | Postoperatively, minimum 2.5 year follow-up
  Secondary outcomes for aim 2: EQ-5D is a five-item instrument to assess health status in the following five dimensions: mobility, self-care, usual activity, pain or discomfort, and anxiety or depression. Individual domain scores will be converted to a summary index representing utility weights, which allow conduct of cost-effectiveness analyses.
Mental and physical health symptoms according to PROMIS instruments | Postoperatively, minimum 2.5 year follow-up
  Secondary outcomes for aim 2: Physical and mental health symptoms and physical functioning will be measured with standardized PROMIS instruments, including: Pain interference, Neuropathic Pain, Fatigue, Sleep disturbance, Depression, Anxiety, and Physical Function. A mean of 50 and a standard deviation of 10 represent the general population in the US.

OTHER OUTCOMES:
Other recorded outcomes (safety endpoints) | Within 30 days of surgery or during index hospitalization, whichever is longer.
  30-day mortality and major postoperative complications (revision for bleeding, perioperative MI (<48 hours after surgery), need for dialysis, need for tracheostomy, and surgical site complications).

CONTACTS AND LOCATIONS:
Overall Officials: Mario Gaudino, Prof/PhD/MD, Principal Investigator — Weill Medical College of Cornell University; Stephen Fremes, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Ruth Masterson Creber, RN, PhD, Principal Investigator — Columbia University; C. Noel Bairey Merz, MD, Principal Investigator — Cedars-Sinai; Karla Ballman, PhD, Principal Investigator — Weill Medical College of Cornell University; Sean O'Brien, PhD, Principal Investigator — Duke University
Locations (141):
- United States (41):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale University Hospital, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Baystate Health, Springfield, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Nebraska Heart Hospital, Lincoln, Nebraska
  - Methodist Physicians Health, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Englewood Health, Englewood, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - NewYork-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Weill Cornell Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - New York Presbyterian Queens, Queens, New York
  - Duke University, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Genesis Healthcare System, Zanesville, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Baylor Scott & White Research Institute, Dallas, Texas
  - The University of Texas Medical Health Branch at Galveston, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - UT Health San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
- Australia (2):
  - Victorian Heart Hospital, Clayton
  - The University of Melbourne, Melbourne
- Austria (5):
  - Medical University of Graz, Graz
  - Innsbruck Medical University, Innsbruck
  - Kepler University Hospital, Linz
  - Medical University of Vienna, Vienna
  - Krankenhaus Nord Vienna North Hospital, Vienna
- Brazil (3):
  - Institute of Cardiology Porto Alegre, Porto Alegre
  - Heart Institute University of São Paulo, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, Vila Mariana
- Canada (15):
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Horizon Health Network - Saint John Regional Hospital, Saint John, New Brunswick
  - NL Health Services, St. John's, Newfoundland and Labrador
  - Health Sciences North, Greater Sudbury, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - University Hospital of Montreal, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Ste Foy, Quebec
  - Hopital Sacre-Coeur, Montreal
  - Fraser Clinical Trials, New Westminster
- China (4):
  - Fuwai Hospital China, Beijing, Beijing Municipality
  - Jilin Heart Hospital China, Changchun, Jilin
  - Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Teda Hospital Tianjin China, Tianjin, Tianjin Municipality
- University Hospital Dubrava, Zagreb, Croatia
- Czechia (2):
  - University Hradec Králové, Hradec Králové
  - General University Hospital, Prague, New Town
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, Copenhagen
- Germany (14):
  - Universitäts-Herzzentrum Bad Krozingen Freiburg, Bad Krozingen, Baden-Wurttemberg
  - HDZ NRW Bad Oeynhausen Germany, Bad Oeynhausen
  - Deutsches Herzzentrum der Charite, Berlin
  - Duisburg Heart Center, Duisburg
  - Dusseldorf University, Düsseldorf
  - University Hospital Erlangen, Erlangen
  - Essen University, Essen
  - Frankfurt University, Frankfurt
  - University Hospital of Giessen and Marburg, Giessen
  - University Medical Center of Göttingen, Göttingen
  - Jena University Hospital, Jena
  - Heart Center Herzzentrum, Leipzig, Leipzig
  - Robert-Bosch-Hospital Stuttgart Germany, Stuttgart
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
- India (2):
  - G Kuppuswamy Naidu Memorial Hospital (GKNM), Coimbatore, Tamil Nadu
  - Star Hospitals - Hyderabad, India, Hyderabad, Telangana
- Rambam Health Care Campus, Haifa, Israel
- Italy (8):
  - Anthea Hospital, Bari
  - Humanitas Gavazzeni of Bergamo, Bergamo
  - Fondazione Poliambulanza, Brescia
  - Maria Cecilia Hospital GVM, Cotignola
  - Careggi University Hospital, Florence
  - European Hospital, Roma
  - Universita' Cattolica del Sacro Cuore, Roma
  - Ospedale Le Molinette, Torino, Torino
- Japan (2):
  - Tokyo Medical and Dental University, Bunkyō-Ku, Tokyo
  - Saitama Medical University Japan, Saitama
- Netherlands (3):
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - Maastricht University Medical Centre, Maastricht
- Acibadem-Sistina Hospital, Skopje, North Macedonia
- Poland (3):
  - Medical University Gdansk, Gdansk
  - Medical University of Silesia, Katowice
  - Zbigniew Religa Lower Silesian Heart Disease Centre, Zabrze
- Portugal (4):
  - University Hospital Coimbra, Coimbra
  - Centro Hospitalar Lisboa Ocidental, Lisbon
  - Centro Hospitalar e Universitário Sao Joao, Porto
  - Centro Hospitalar e Universitário Sao João, Porto
- National Research Medical Center of the Russian Academy of Sciences - Tomsk, Russia, Tomsk, Russia
- Dedinje Cardiovascular Institute, Belgrade, Serbia
- National University of Singapore, Singapore, Singapore
- South Korea (2):
  - Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul
  - Seoul National University Hospital, Seoul
- Spain (4):
  - Hospital Universitario del Vinalopo, Elche, Alicante
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clinico de San Carlos, Madrid
  - NavarraBiomed, Pamplona
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Karonlinska University Hospital, Stockholm
- National Taiwan University Hospital, Zhongzheng, Taipei, Taiwan
- United Kingdom (16):
  - Blackpool Teaching Hospitals NHS Trust, Blackpool, Lancashire
  - Oxford University Hospitals NHS Trust, Multiple Locations, Oxford
  - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire
  - Royal Papworth NHS Foundation Trust, Cambridge
  - NHS Golden Jubilee, Clydebank
  - The Royal Infirmary of Edinburgh, Edinburgh
  - Hull University Hospitals, Hull
  - University Hospitals of Leicester, Leicester
  - Liverpool Heart and Chest Hospital Foundation Trust, Liverpool
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - St George's University Hospitals, London
  - Manchester University NHS Trust, Manchester
  - South Tees Hospitals NHS Trust, Middlesbrough
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Royal Wolverhampton NHS Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Primary outcome data under request
Supporting Information: Study Protocol, SAP
Time Frame: From publication until the third year after publication
Access Criteria: Research scope

REFERENCES:
- [Background] Loop FD, Lytle BW, Cosgrove DM, Stewart RW, Goormastic M, Williams GW, Golding LA, Gill CC, Taylor PC, Sheldon WC, et al. Influence of the internal-mammary-artery graft on 10-year survival and other cardiac events. N Engl J Med. 1986 Jan 2;314(1):1-6. doi: 10.1056/NEJM198601023140101. PMID 3484393
- [Background] Tatoulis J, Buxton BF, Fuller JA. Patencies of 2127 arterial to coronary conduits over 15 years. Ann Thorac Surg. 2004 Jan;77(1):93-101. doi: 10.1016/s0003-4975(03)01331-6. PMID 14726042
- [Background] Lytle BW, Blackstone EH, Loop FD, Houghtaling PL, Arnold JH, Akhrass R, McCarthy PM, Cosgrove DM. Two internal thoracic artery grafts are better than one. J Thorac Cardiovasc Surg. 1999 May;117(5):855-72. doi: 10.1016/S0022-5223(99)70365-X. PMID 10220677
- [Background] Taggart DP, D'Amico R, Altman DG. Effect of arterial revascularisation on survival: a systematic review of studies comparing bilateral and single internal mammary arteries. Lancet. 2001 Sep 15;358(9285):870-5. doi: 10.1016/S0140-6736(01)06069-X. PMID 11567701
- [Background] Yi G, Shine B, Rehman SM, Altman DG, Taggart DP. Effect of bilateral internal mammary artery grafts on long-term survival: a meta-analysis approach. Circulation. 2014 Aug 12;130(7):539-45. doi: 10.1161/CIRCULATIONAHA.113.004255. Epub 2014 Jun 10. PMID 24916209
- [Background] Hillis LD, Smith PK, Anderson JL, Bittl JA, Bridges CR, Byrne JG, Cigarroa JE, Disesa VJ, Hiratzka LF, Hutter AM Jr, Jessen ME, Keeley EC, Lahey SJ, Lange RA, London MJ, Mack MJ, Patel MR, Puskas JD, Sabik JF, Selnes O, Shahian DM, Trost JC, Winniford MD; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; American Association for Thoracic Surgery; Society of Cardiovascular Anesthesiologists; Society of Thoracic Surgeons. 2011 ACCF/AHA Guideline for Coronary Artery Bypass Graft Surgery. A report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Developed in collaboration with the American Association for Thoracic Surgery, Society of Cardiovascular Anesthesiologists, and Society of Thoracic Surgeons. J Am Coll Cardiol. 2011 Dec 6;58(24):e123-210. doi: 10.1016/j.jacc.2011.08.009. Epub 2011 Nov 7. No abstract available. PMID 22070836
- [Background] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Background] Aldea GS, Bakaeen FG, Pal J, Fremes S, Head SJ, Sabik J, Rosengart T, Kappetein AP, Thourani VH, Firestone S, Mitchell JD; Society of Thoracic Surgeons. The Society of Thoracic Surgeons Clinical Practice Guidelines on Arterial Conduits for Coronary Artery Bypass Grafting. Ann Thorac Surg. 2016 Feb;101(2):801-9. doi: 10.1016/j.athoracsur.2015.09.100. Epub 2015 Dec 8. PMID 26680310
- [Background] Benedetto U, Raja SG, Albanese A, Amrani M, Biondi-Zoccai G, Frati G. Searching for the second best graft for coronary artery bypass surgery: a network meta-analysis of randomized controlled trialsdagger. Eur J Cardiothorac Surg. 2015 Jan;47(1):59-65; discussion 65. doi: 10.1093/ejcts/ezu111. Epub 2014 Mar 30. PMID 24686003